CLINICAL TRIAL: NCT01442272
Title: Clinical Trial, Open, Parallel Groups , Value the Antiproteinuric Effects From Vitamin D Derivatives in Patient With Chronic Kidney Illness and the Lack of Vitamin D
Brief Title: Value Antiproteinuric Effects From Vitamin D Derivatives in Patient With Chronic Kidney Illness and the Lack of Vitamin D
Acronym: NEFROVID2010
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario de Canarias (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEFROVID2010
Record Dates: First submitted 2011-09-26; First posted 2011-09-28 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2011-09

CONDITIONS: Kidney Failure, Chronic; Disorder of Vitamin D
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Calcifediol; paricalcitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Habitual medication withuot additional (No Intervention)
  Interventions: Drug: Habitual medication
- Habitual medication plus Hidroferol® (Active Comparator)
  Interventions: Drug: Hidroferol®
- Habitual medication plus Zemplar® (Active Comparator)
  Interventions: Drug: Paricalcitol: Zemplar®

INTERVENTIONS:
Drug: Hidroferol® — Hidroferol® drinkable ampoule in oral solution, 266 mcg (1 drinkable ampoule) each 15 days during 12 months
  Other Names: B
  Arms: Habitual medication plus Hidroferol®
Drug: Paricalcitol: Zemplar® — Paricalcitol (Zemplar®) oral capsule , 1 mcg (1 capsule)each 24 hours during 12 months
  Other Names: C
  Arms: Habitual medication plus Zemplar®
Drug: Habitual medication — Habitual medication
  Other Names: A
  Arms: Habitual medication withuot additional

SUMMARY:
The purpose of this study is to determine the value the additional antiproteinuric effects of vitamin D derivatives treatment, in patients with Chronic Kidney Illness phase II-IV, with lack of vitamin D and residual proteinuria higher 0,5 grams/day.

ELIGIBILITY:
Inclusion Criteria:

* Male/female Patients older 18 years old
* Patients have signed written informed consent
* Chronic Kidney Illness phase II-IV plus residual proteinuria >0,5 grams/day (two or more consecutive occasions) and plus beta blockers treatment from AARS during al least 3 months.
* Serum levels of calcifediol in the lack of level (15-30 ng/ml).

Exclusion Criteria:

* Bad control of high blood pressure (higher or same 180/110 mmHg)
* Bad control of diabetes (HbA1c higher 9,5 in the last three months period)
* Hypercalcemia (<10,2 mg/dL) o hyperphosphatemia(>5,5 mg/dL), CaxPO4>50, hypercalciuria (urin Ca/Cr quotient > 0,15)
* Vitamin D treatment or any analogous
* Hepatic failure ( AST o ALT > 3 times higher than normal limit)
* medical history of poor nutrient intestinal absorptions or chronic diarrhea
* Active nephrolithiasis
* Treatment with medication wich can change vitamin D metabolism (phenobarbital, phenytoin, rifampicin)
* Participation in other Clinic Trial in 3 last months
* Active Alcoholism
* Neoplasia precedent (except cutaneous no melanoma)
* Pregnant women or while breastfeeding
* Vitamin D hypersensitivity or any its excipient hypersensitivity
* Any other condition from Research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Protein/creatinine quotient and albumin/creatinine in matinal urine sample: basal and 3 period months after a month of the therapeutic protocol beginning. | 1-3 month

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, S/C Tenerife
  - HUC, San Cristóbal de La Laguna, S/c Tenerife